CLINICAL TRIAL: NCT00589433
Title: Follow Up Study of Tear in the Rotator Culf
Status: Terminated | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Evaluation of the rotator cuff tear using Ultra sound, Hadassah Medical Organization
Other Study IDs: SAF02-HMO-CTIL
Record Dates: First submitted 2008-01-01; First posted 2008-01-09 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Rotator Culf Tear

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Rotator culf tears are common in the aging population and are a significant morbidity source. The common knowledge is that the major tears do not heal and constantly expanding.Still since the majority of the patients are old the acceptable therapy is conservative treatment.

Our objective is to estimate the accuracy of rotator culf tear utilizing an ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Was diagnosed with shoulder tear
* Size of the tear till 2.5 cm
* The opposite tendon-normal

Exclusion Criteria:

* systematic Diseases .
* Injury to the shoulder after the previous US.
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Safran, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Orthopedic Department, Jerusalem, Israel